CLINICAL TRIAL: NCT00514969
Title: Protein-Tyrosine Kinase Inhibitor (STI571) for Treatment of Patients With Ph+ Chronic Myeloid Leukemia in Accelerated and Blastic Phase. A Phase II Study
Brief Title: Protein-Tyrosine Kinase Inhibitor (STI571) for Treatment of Patients With Ph+ Chronic Myeloid Leukemia in Accelerated and Blastic Phase
Acronym: CML003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML003
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Myeloid Leukemia
Keywords: accelerated and blastic phase; STI571
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib (STI571)

SUMMARY:
This is a phase II, multi-center, open-label, non-randomized trial. During Part 1 of the trial, patients will receive once daily oral administration of STI571 at a dose of 600 mg for 24 weeks. After completing 24 weeks of therapy, patients may be eligible to receive additional therapy during Part 2 of the trial provided that, in the opinion of the investigator, the patient has benefited from treatment with STI571 and in the absence of safety concerns. During Part 2 (which is of indefinite duration), patients will continue to receive STI571 on a daily basis until either death, the development of intolerable toxicity or the investigator feels it is no longer in the patient's best interest to continue therapy, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients * 18 years of age
2. Accelerated phase of CML defined as the presence of one or more of the following:

   * percentage of blasts in blood or bone marrow * 15% but < 30%
   * percentage of blasts plus promyelocytes in the peripheral blood or bone marrow * 30% (providing that < 30% blasts are present in the bone marrow)
   * peripheral basophils * 20%
   * thrombocytopenia < 100 x 109/L unrelated to therapy These criteria must be met within 4 weeks of administration of first dose of trial treatment.
3. Blastic phase of CML defined as the presence of one or more of the following:

   * percentage of blasts in blood or bone marrow * 30%
   * percentage of blasts and promyelocytes in blood or bone marrow * 50%
   * documented extramedullary blast involvement (skin, lymph node, bone, lung).
4. Voluntary written informed consent.

Exclusion Criteria:

1. Patients of childbearing potential wihout a negative pregnancy test prior to the initiation of study drug. Barrier contraceptive precautions are to be used throughout the trial in both sexes.
2. Patients with an ECOG Performance Status Score ** 3 (see Section 7.2.1)
3. Creatinine levels more than 2 x's the ULN at the laboratory where the analysis was performed.
4. Total serum bilirubin more than 1.5 x's the upper limit of the normal range (ULN) at the laboratory where the analyses were performed; in patients with clinically suspected leukemic involvement of the liver, total bilirubin more than 3 x's the ULN
5. AST (SGOT) or ALT (SGPT) more than 3 x's the upper limit of the normal range (ULN) at the laboratory where the analyses were performed; in patients with clinically suspected leukemic involvement of the liver, AST and ALT more than 5 x's the ULN
6. Patients receiving treatment with interferon-alpha within 48 hours of Day 1.
7. Patients receiving treatment with hydroxyurea within 24 hours of Day 1
8. Patients receiving treatment with homoharringtonine within 14 days of Day 1
9. Patients receiving treatment with low-dose cytosine arabinoside (< 30 mg/m2 every 12 to 24 hours administered daily) within seven days of Day 1
10. Patients receiving treatment with moderate dose cytosine arabinoside (100-200 mg/m2 for 5 to 6 days) within 14 days of Day 1.
11. Patients receiving treatment with high-dose cytosine arabinoside (1-3 g(m2 every 12 to 24 hours for six to 12 doses) within 28 days of Day 1.
12. Patients receiving anthracyclines, mitoxantrone, etoposide, methotrexate or cyclophosphamide within 21 days of Day1.
13. Patients receiving busulfan within six weeks of Day 1.
14. Patients receiving anti-leukemic agents not included in Exclusion Criteria 6-13 should not begin treatment with STI571 until sufficient time has elapsed for potential recovery to have occurred in the nadir in blood counts. In practice, a full recovery of blood counts may not be possible due to progression of the underlying disease.
15. Patients receiving any hematopoietic stem cell transplantation and who have not achieved full hematopoietic recovery following the transplant
16. Patients receiving any other investigational agents within 28 days of Day 1.
17. Patients with Grade ¾ cardiac disease.
18. Patients with any serious concomitant medical condition
19. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.
20. Patients with a prior diagnosis of accelerated or blastic phase who are in remission and do not fit inclusion criteria, are not eligible.
21. Patients who are likely to be submitted to any procedure of stem cell transplantation before the end of the treatment (6 months), are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

PRIMARY OUTCOMES:
To determine the rate of hematological response lasting * 4 weeks in adult patients with Ph chromosome positive CML in accelerated and blastic phase

SECONDARY OUTCOMES:
duration of hematological response and overall survival, cytogenetic response and safety

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli" Università degli Studi di Bologna
Locations (1):
- Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli" Università degli Studi di Bologna, Bologna, Italy

REFERENCES:
- [Derived] Palandri F, Castagnetti F, Testoni N, Luatti S, Marzocchi G, Bassi S, Breccia M, Alimena G, Pungolino E, Rege-Cambrin G, Varaldo R, Miglino M, Specchia G, Zuffa E, Ferrara F, Bocchia M, Saglio G, Pane F, Alberti D, Martinelli G, Baccarani M, Rosti G; GIMEMA Working Party on Chronic Myeloid Leukemia. Chronic myeloid leukemia in blast crisis treated with imatinib 600 mg: outcome of the patients alive after a 6-year follow-up. Haematologica. 2008 Dec;93(12):1792-6. doi: 10.3324/haematol.13068. Epub 2008 Oct 6. PMID 18838477